CLINICAL TRIAL: NCT05828992
Title: Benchmarking Integrated Care for People Living With Huntington's Disease in England (Integrate-HD Study)
Brief Title: Benchmarking Integrated Care for People Living With Huntington's Disease in England
Acronym: Integrate-HD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Central Coast Research Institute for Integrated Care, Australia (Unknown); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ERGO number: 77725
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Huntington Disease
Keywords: Integrated care; Huntington's Disease; Caregiver; Person-centred care; Benchmarking; Survey
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Person at risk: Survey personalised for people living at risk of developing Huntington's Disease, meaning they have a parent diagnosed with HD but the person themselves have not undertaken a genetic test.
  Interventions: Other: No intervention administered
- Person HD gene positive asymptomatic: Survey personalised for people that tested positive in their predictive genetic test but have not been yet diagnosed with clinical HD (manifest HD).
  Interventions: Other: No intervention administered
- Person HD gene positive symptomatic: Survey personalised for people that tested positive in their predictive genetic test and have been diagnosed with clinical HD (manifest HD).
  Interventions: Other: No intervention administered
- Informal caregiver: Survey personalised for people caring for another person diagnosed with HD.
  Interventions: Other: No intervention administered
- Former informal caregiver: Survey personalised for people that have cared for another person diagnosed with HD in the last 3 years.
  Interventions: Other: No intervention administered

INTERVENTIONS:
Other: No intervention administered — Survey only to gather people's experiences, opinions and needs.

SUMMARY:
The survey and full study information can be accessed here: https://southampton.qualtrics.com/jfe/form/SV_8iEedDJZy4xaiI6

The goal of this anonymous survey is to benchmark integrated care from the perspective of service users in adults living with Huntington's Disease, including informal caregivers. The main question it aims to answer is: Is standard of care for people living with HD in England person-centred integrated care from the perspective of service users?

Participants will complete a one-time anonymous survey either online or on paper, according to their preference, that takes an average of 20-30 minutes. Participants can take breaks as needed, picking up the survey from where it was paused.

DETAILED DESCRIPTION:
Huntington's disease (HD) is a rare brain disease that affects people's coordination, thinking and behaviour. It is a hereditary condition, affecting families across generations. Because its complex, it requires different sectors working together. Different surveys can be found in long term neurological conditions indicating care fragmentation and unmet severe needs, but evidence in HD is sparse.

Two surveys were identified covering people's needs in the UK, dated from 2006 and 2010. When looking for models or approaches tested to improve outcomes for people living with HD, no studies were found. This is an underserved population with complex needs and care gaps that remain unaddressed.

Little is known about to what extent people living with HD are experiencing care coordination between services and sectors in England. Integrate-HD aims to find out what good, joined-up care looks like. The study will explore the views and experiences of people living with HD, to identify the changes needed to improve people's care and quality of life.

Integrate-HD is a national survey to benchmark integrated care from the perspective of people living with HD, including informal caregivers.

The study objectives are to:

1. Characterise and classify systems/organisations in England involved in HD care in relation to person-centred integrated care from the perspective of users.
2. Identify areas considered integrated by service users.
3. Identify areas considered fragmented by service users.
4. Map care resources used by people living with HD in England.
5. Identify unmet care needs that need improvement.

ELIGIBILITY:
Inclusion Criteria:

Adults with capacity living in England and fluent in English that are:

* A person at risk of HD (where at least one parent is diagnosed with HD, therefore their offspring has 50% chance of developing the disease);
* A person diagnosed with HD symptomatic or asymptomatic (after undergoing gene testing and having a positive result);
* An informal caregiver supporting someone living with HD;
* A former informal caregiver with experience of supporting someone living with HD in the last 3 years.

Exclusion Criteria:

* Below 18 years old;
* Not fluent in English;
* A person without capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with capacity living in England impacted by Huntington's Disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Level of integration | 9 months
  Using SPSS (version 27) responses will be analysed to explore the level of integration at specific systems or organizations in England to distinguish between "higher" and "lower" integration levels. The Likert-type scale section of the survey will have a scheme of points attributed to generate a key of integration level per domain.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra B Pires, MSc, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
During this study all information collected from participants will be kept confidential. The data gathered through surveys is anonymous and will be stored on a secure database using only survey IDs. Any identifiable information, such as email contact provided at the end of the survey (in order to receive updates on the research or show interest in future research) will be stored separately to survey answers.
  All data will be stored on a password protected university computer/laptop or in a locked filing cabinet in a secure office in the University. This will only be accessible by the research team. The procedures for handling, processing, storing, and destroying data are compliant with the Data Protection Act 2018.